CLINICAL TRIAL: NCT04494737
Title: A Neuroscientific Account of Embodied Ethics: Mindfulness Training Related Improvements In Moral Reasoning
Brief Title: Wellbeing, Stress Reduction and Social Cognition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Sara W Lazar, Associate Researcher in Psychiatry, Assistant Professor in Psychology, Massachusetts General Hospital
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 2020A001098
Record Dates: First submitted 2020-02-14; First posted 2020-07-31 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Cognitive Function 1, Social

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Comparator: Program 1 (Active Comparator): Mindfulness Training program is based on mindfulness based stress reduction developed by Kabat-Zinn, but the didactic content is focused on attention training and meta-awareness. Participants will be taught formal open awareness meditation, gentle yoga, and a 'body scan' meditation during weekly classes. Importantly, there is no retreat day included in the program.
  Interventions: Behavioral: Active Comparator: Program 1
- Active Comparator: Program 2 (Active Comparator): Stress Management Education (SME) is designed to control for non-specific factors such as contact hours, stress education, and gentle exercise. Stress education classes will consist of teaching about the effects of stress on health and optimizing one's personal health care, understanding positive coping behavior, optimizing nutrition to decrease stress, and exercise and strength training.
  Interventions: Behavioral: Active Comparator: Program 2

INTERVENTIONS:
Behavioral: Active Comparator: Program 1 — A well-established behavioral method for reducing stress. To maintain blinding, details will be given to participants after randomization.
  Arms: Active Comparator: Program 1
Behavioral: Active Comparator: Program 2 — A well-established behavioral method for reducing stress. To maintain blinding, details will be given to participants after randomization.
  Arms: Active Comparator: Program 2

SUMMARY:
There are many ways to improve wellbeing. This study will compare two 8-week wellbeing training programs. In addition to looking at how well the programs reduce stress and enhance wellbeing, the investigators will also ask questions about how these programs influence cognition and decision making.

DETAILED DESCRIPTION:
The training programs that aim to reduce stress and enhance wellbeing differ in terms of the techniques they utilize, as well as in terms of their mechanisms of change. These different mechanisms may have different impact on cognition and decision making. The aim of the study is to compare the different programs and also explore potential mediators of changes in wellbeing.

ELIGIBILITY:
Inclusion Criteria:

1. 18-65 years of age.
2. Right-handed.
3. Able to speak, understand, and read English.
4. Willing to participate in a 20-week study period and undergo 2 MRI scans at Massachusetts General Hospital (MGH).
5. Able to safely undergo an MRI scan.
6. Stable medication/treatment regimen (changes in medication must have occurred three months prior to enrollment in this study).
7. Subjects with well-controlled vascular risk factors, such as treated hypertension, treated hyperlipidemia or well-controlled Type II diabetes (glucose levels < 250) will be included.
8. Subjects with a history of cerebrovascular problems but have no persistent neurological deficits will be included.
9. Available for scheduled class times for both study courses.
10. Will be staying in the study area for the next 3 months.
11. Able to complete up to 40 minutes of homework per day during the 8-week course.

Exclusion Criteria:

1. Cardiovascular disease, stroke, or congestive heart failure.
2. Has any of, or is; surgical aneurysm clips, neurostimulator, implanted pumps, metal fragments in eyes, pregnant, cardiac pacemaker, non-removable nitroglycerin patch, non-MRI compatible cochlear implants, any other non-MRI compatible metal in body.
3. Has permanent bridgework in upper mouth that could interfere with MRI scan.
4. Active hematological, renal, pulmonary, endocrine or hepatic disorders.
5. A history of neurological disease or injury, including a history of seizures or significant head trauma (i.e., extended loss of consciousness, bleeding in the brain, Parkinson's disease, stroke).
6. Received treatment for cancer within the last year (skin cancer will be allowed as will any cancer more than 2 years since the last treatment).
7. Diagnosis of schizophrenia, post traumatic stress disorder (PTSD), bipolar disorder, or psychotic disorder at any point during lifetime.
8. Diagnosis of any axis I psychiatric disorder within the last 12 months.
9. Weighs more than 350 pounds
10. Neurological or medical conditions that would interfere with study procedures or confound results, such as conditions that alter cerebral blood flow or metabolism.
11. Unstable medications or on medications with CNS effects including cholinesterase inhibitors, memantine and antidepressants.
12. Use of psychotropic medications within 12 months prior to study.
13. Daily use of any medication that alters neural metabolism or blood flow, including chronic use of benzodiazepines, potent central nervous system (CNS) penetrant anticholinergic medications (for bladder control or allergies). These medications taken on an as needed basis (prn) will be allowed. (Over the counter supplements, such as Gingko and fish oil will be allowed.)
14. Any other medications as reviewed by a clinician on a case-by-case basis.
15. Current regular formal practice of meditation, tai chi, Feldenkrais or other mind-body practice with a teacher for more than 2 months within the past year, or more than 1 year of practice within the last 10 years. Significant prior mind-body experience as determined by the PI based on frequency, duration, recency and type of practice.
16. Has claustrophobia.
17. Any other criteria that will interfere with the subject's participation as determined by a study doctor.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-01-05 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Neural functioning during moral decision-making | baseline, week 8
  The name of the measurement is neural functioning during moral decision-making. To assess neural functioning, participants will undergo a functional MRI scan while they perform a moral judgment task. The task that involves moral (n=18) and non-moral (n=18) dilemma vignettes. These dilemmas have been validated and will be presented as text in an event related design. The participant specific task-related brain activity will be generated by contrasting brain activity between moral and non-moral dilemmas using Statistical Parametric Mapping software. The unit of measure is BOLD signal and the blood-oxygen level dependent (BOLD) signal contrast of interest is moral vs. nonmoral dilemmas.

SECONDARY OUTCOMES:
Moral Reasoning Ability | baseline, week 8, week 16
  Defining Issues Test-2 (DIT-2) is the name of the measurement. It is a survey, that assesses participants' developmental level of moral reasoning ability. The resulting scores at the DIT-2 test indicate levels of higher order moral reasoning.

CONTACTS AND LOCATIONS:
Overall Officials: Gunes Sevinc, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- MGH, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No